CLINICAL TRIAL: NCT00126672
Title: A Phase II Multi-Center Study of Rapamycin for Treating Kidney Angiomyolipomas in TSC or LAM Patients
Brief Title: RAPAMYCIN FOR KIDNEY ANGIOMYOLIPOMAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Tuberous Sclerosis Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-298; R01CA107164 (NIH); P30CA006516 (NIH)
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Nonmalignant Neoplasm; Tuberous Sclerosis; Lymphangioleimyomatosis; Kidney Angiomyolipoma
Keywords: angiomyolipoma
MeSH Terms: conditions — Neoplasms; Tuberous Sclerosis; Angiomyolipoma | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ramaycin (Experimental): Rapamycin treatment was initiated with a loading dose of 6 mg by mouth on day 1 followed by 2 mg by mouth daily. The dose was then adjusted to maintain a target blood level of 3-9 ng/ml for the first 16 weeks. After week 16, the dose of Rapamycin was increased to a target level of 9-15 ng/ml unless there was evidence for a partial response or complete response by kidney MRI. Trough Rapamycin levels were checked every 8-12 weeks (at 24 weeks, 32 weeks, 40 weeks, and 52 weeks) in all patients until the 12-month (week 52) study visit. If the Rapamycin dose was below target, the dose was increased by 1-2 mg until the target trough level was achieved. Rapamycin levels were checked every 2-3 weeks while the dose was adjusted. Amendment 20 (Jan 2009) permitted additional Rapamycin treatment during months 12-24 if the treating site investigator judged that this was in the best interest of the study participant.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin
  Other Names: Rapamune; Sirolimus

SUMMARY:
This research study is evaluating a drug called rapamycin as a possible treatment for the lumps (or tumors) that form in the kidneys, called angiomyolipomas, in people who have either TSC or LAM. Kidney angiomyolipomas are tumors that are made up of blood vessels, muscle and fat. Rapamycin has been approved to treat other diseases, but it is investigational for treating kidney angiomyolipomas.

Investigational means that it is being as a possible treatment for kidney angiomyolipomas but is not currently approved by the U.S. Food and Drug Administration (FDA) for treating this disease.

DETAILED DESCRIPTION:
This research study is a Phase ll clinical trial. Phase II clinical trials test the effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it-such as the safest dose to use, the side effects it may cause, and if the drug is effective for treating different types of diseases. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved this drug for this type of disease.

The purpose of this research study is to see if the drug, rapamycin, is effective in treating kidney angiomyolipomas. Rapamycin is a drug that may decrease the size of tumors. This drug has been used in treating other diseases and cancers in humans and information from those other research studies suggests that rapamycin may help to shrink tumors in this research study.

The investigators will also be looking at the safety of this drug in people with TSC or LAM. In addition, the investigators will also look at whether this drug is effective for treating other conditions that occur in people that have TSC or LAM (tubers, subependymal giant cell astrocytomos, facial angiofibromas, kidney cysts in TSC, or symptoms of cough, breathing trouble or other symptoms of lung problems in people with LAM).

Although these tumors (kidney angiomyolipomas) may not change for many years, they do not go away on their own. They often grow larger and may bleed. The standard of care for treating these tumors is to take pictures of them using ultrasound, CT or MRI (called kidney imaging) every 1-3 years to see if they are getting larger or if they are bleeding. If they do grow larger or bleed, removing them by surgery or cutting off the blood supply to the tumor (vascular embolization) may be recommended.

This research study is being done because there are no medicines available at this time that can treat kidney angiomyolipomas. However, recent studies in the laboratory have shown that the drug, rapamycin, maybe effective in treating these tumors. Because rapamycin is approved by the FDA for treating other medical conditions, we know what doses are safe to use based on guidelines that have been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-65 years old (females of reproductive age must not be pregnant or breastfeeding)
* Kidney ANGIOMYOLIPOMA 2 cm or greater on baseline MRI (a CT scan may be used for patients who cannot undergo MRI imaging)
* No evidence of severe LAM (not on continuous oxygen)
* Informed consent, including consent for submission of blood, urine and tissue samples as described in the appendix.
* Adequate renal and liver function (eGFR of 30 or higher, SGOT, SGPT, TBili, Alk Phos all<2x normal)
* HCT>27%
* ANC > 1500 and platelet count >100,000
* Diagnosis of TSC or LAM (diagnosis of TSC using revised diagnostic criteria [45], diagnosis of LAM made by chest CT scan and reviewed by a pulmonologist).
* Fertility/Reproductive issues: The effects of rapamycin on the developing fetus at the doses used in this study are unknown. For this reason, rapamycin should not be taken during pregnancy. Participants who are fertile must maintain adequate contraception while they are taking rapamycin and for twelve weeks after stopping the drug. Acceptable contraceptive measures include prior hysterectomy, oophorectomy or tubal ligation, complete abstinence, barrier methods which include both a cervical diaphragm and spermicidal jelly, and progestin based contraceptives. Pregnancy tests will be obtained at enrollment and during study visits at 8 weeks, 16 weeks, 24 weeks, 32 weeks, 40 weeks, and 52 weeks.

  * Note: Eligibility requirement of ECOG PS of 0 or 1 has been removed to allow participation of those subjects with TSC who are classified as ECOG PS of 2,3, or 4 because of cognitive impairment rather than progressive disease. This change allows site Pl's to individualize decision making on whether or not to enroll such subjects after discussing details of the study with prospective participant and legal guardian. The decision to enroll individuals with ECOG PS of 2,3, or 4 will be at the discretion of the Principal Investigator.

Exclusion criteria:

* Unstable seizures (defined as changes in anti-epileptics OR increase in frequency and/or severity or seizures in the 60 days prior to study entry)
* Significant bleed associated with kidney angiomyolipoma(s) (defined as bleed associated with shock OR requiring a blood transfusion in the 30 days prior to study entry)
* Severe LAM (defined as dependent on continuous supplemental oxygen)
* Evidence for accelerating renal dysfunction or acute renal failure
* Diagnosis of Renal Cell Cancer that has not been treated (additional clarification: individuals with a prior history of renal cancer who have had appropriate surgery and have no evidence of metastatic disease can be enrolled)
* Active infection
* Patients will be excluded if they have been treated with any investigational agent in the 30 days prior to study entry
* Patients may not be treated with other investigational agents while on study
* Prior history of coronary artery disease
* Vascular embolization for treatment of kidney angiomyolipoma(s) within 6 months
* Patients who must take diltiazem, ketoconazole or rifampin chronically will be excluded because of known drug interactions. Both diltiazem and ketoconazole are strong inhibitors of CYP3A4 and are known to increase rapamycin levels. Rifampin is a known CYP3A4 and P-glycoprotein inducer and is known to significantly reduce rapamycin levels.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-12-20 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Dabora, MD, PhD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (7):
- United States (7):
  - Loma Linda University School of Medicine, Loma Linda, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malinowska IA, Lee N, Kumar V, Thiele EA, Franz DN, Ashwal S, Sagalowsky A, Dimario FJ Jr, Cutler D, Krueger D, Camposano S, Paolini J, Dabora SL. Similar trends in serum VEGF-D levels and kidney angiomyolipoma responses with longer duration sirolimus treatment in adults with tuberous sclerosis. PLoS One. 2013;8(2):e56199. doi: 10.1371/journal.pone.0056199. Epub 2013 Feb 20. PMID 23437092
- [Derived] Dabora SL, Franz DN, Ashwal S, Sagalowsky A, DiMario FJ Jr, Miles D, Cutler D, Krueger D, Uppot RN, Rabenou R, Camposano S, Paolini J, Fennessy F, Lee N, Woodrum C, Manola J, Garber J, Thiele EA. Multicenter phase 2 trial of sirolimus for tuberous sclerosis: kidney angiomyolipomas and other tumors regress and VEGF- D levels decrease. PLoS One. 2011;6(9):e23379. doi: 10.1371/journal.pone.0023379. Epub 2011 Sep 6. PMID 21915260

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapamycin: After the screening procedures confirm that you are eligible to participate in the research study
  * Rapamycin: oral, 3-9 ng/ml daily for 4 months, then increase dose to 9-15 ng/ml for 20 months.
  * MRI/CT scan at 16 week, 32 weeks, 52 weeks during treatments.
Period: Overall Study
Arm/Group | Rapamycin
Started | 36
Completed | 28
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Ramaycin: After the screening procedures confirm that you are eligible to participate in the research study
  * Rapamycin: oral, 3-9 ng/ml daily for 4 months, then increase dose to 9-15 ng/ml for 20 months.
  * MRI/CT scan at 16 week, 32 weeks, 52 weeks during treatments.
Arm/Group | Ramaycin
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 34 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34
  Black | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: On treatment, patients were evaluated radiologically for response to therapy up to 52 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramaycin
Number analyzed (Participants) | 36
percentage of participants | 44.4 [28 to 61]

2. Secondary Outcome: Number of Participants With Grade 3 or More Treatment-Related Lymphopenia
Description: All participants reporting maximum grade 3 or more lymphopenia adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv3 on case report forms were counted.
Time Frame: Assessed on treatment up to 52 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramaycin
Number analyzed (Participants) | 36
Participants | 1

3. Secondary Outcome: Number of Participants With no Change Are Observed Changes That Occur in Other TSC Lesions
Description: TSC lesions are tubers, subependymal giant cell astrocytomas, facial angiofibromas, kidney cysts.
Time Frame: Data collected at week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Ramaycin
Number analyzed (Participants) | 36
Participants | 0

ADVERSE EVENTS:
Time Frame: Assessed at 16, 32 and 52 weeks and up to day 30 post-treatment. Treatment duration average (including first 52 weeks) was 78 weeks, range 60-100 weeks.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Ramaycin
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 36/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramaycin (N=36)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 32
Platelet count decreased (Investigations) | 5
White blood cell decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramaycin (N=36)
Anemia (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Jejunal hemorrhage (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 36
Nausea (Gastrointestinal disorders) | 13
Oral pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 26
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
Pain (General disorders) | 4
Allergic reaction (Immune system disorders) | 1
Lung infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 3
Investigations - Other, specify (Investigations) | 3
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 36
Platelet count decreased (Investigations) | 22
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Brachial plexopathy (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 11
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-01-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT00126672/Prot_SAP_000.pdf